CLINICAL TRIAL: NCT03907449
Title: Preview Rapid Strep A Test Method Comparison Study
Status: Suspended | Type: Observational
Why Stopped: Recruitment rates reduced during non-Strep season
Sponsor: Guangzhou Wondfo Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: MDC_2018_Wondfo
Record Dates: First submitted 2019-04-05; First posted 2019-04-09 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Strep Throat

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Symptoms of Strep Throat: Any patient presenting with symptoms of pharyngitis
  * Fever
  * Sore throat
  * Swollen lymph nodes in neck
  * Redness of throat/tonsils
  * White/yellow patches on tonsils
  * Not currently on antibiotics
  Interventions: Diagnostic Test: Preview Rapid Strep A test

INTERVENTIONS:
Diagnostic Test: Preview Rapid Strep A test — Rapid assay for the detection of type A streptococcal infection of the throat.

SUMMARY:
This study is designed to determine the accuracy of the Preview Rapid Strep A Test compared to a laboratory reference method for Group A Streptococcal infection and to determine the precision of the Preview Rapid Strep A test.

ELIGIBILITY:
Inclusion Criteria:

* Any patient presenting with symptoms of pharyngitis

  * Fever
  * Sore throat
  * Swollen lymph nodes in neck
  * Redness of throat/tonsils
  * White/yellow patches on tonsils
  * Not currently on antibiotics
* ≥3 years or older
* Ability to read, understand and sign a consent form, in English, or for parent(s) to sign an assent form providing permission to include children under the age of 18.

Exclusion Criteria:

* Currently taking antibiotics
* Previously enrolled in this study

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 320 patients to be tested, expecting 50-100 positive for Strep A collected from patients of any age and gender from two CLIA waived or waivable sites. Children will be enrolled in this study due to the high prevalence of Strep A infections in minors and the intention to market this investigational device for use for all ages following FDA clearance.
Sampling Method: Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Preview Strep A Rapid Test | 3 months
  Determination of Positive Predictive Value and Negative Predictive Value for Preview Strep A

CONTACTS AND LOCATIONS:
Overall Officials: Paul Granato, PhD, Principal Investigator — UHSH Microbiology; Jagmohan Sidhu, MD, Principal Investigator — UHSH Microbiology
Locations (2):
- United States (2):
  - UHSH Microbiology, Johnson City, New York
  - Summerwood Pediatrics, Liverpool, New York

IPD SHARING:
Plan to Share IPD: No